CLINICAL TRIAL: NCT04555941
Title: Cognitive Effects of Theta Burst Stimulation in Mild Cognitive Impairment and Alzheimer's Disease
Brief Title: The Effects of Intermittent Theta Burst Stimulation in MCI and Early AD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Principal Investigator, Cheng-Chang Yang, Medical researcher, Taipei Medical University Shuang Ho Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: N202003022
Record Dates: First submitted 2020-08-25; First posted 2020-09-21 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Mild Cognitive Impairment; Alzheimer Disease; Cognitive Decline
Keywords: Transcranial magnetic stimulation; non-invasive brain stimulation
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participant and principal investigator do not know what treatment is applied. The outcomes assessor will also be blinded. Only the co-PI who perform the TMS will know the stimulation condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active iTBS (Experimental): The patient is treated with iTBS stimulation according to protocol with an active coil.
  Interventions: Device: intermittent theta burst stimulation
- Sham iTBS (Sham Comparator): The patient is treated with Sham-iTBS stimulation according to protocol with an inactive coil.
  Interventions: Device: intermittent theta burst stimulation

INTERVENTIONS:
Device: intermittent theta burst stimulation — active or Sham iTBS will be given to the AD/MCI patient
  Other Names: Magstim rapid 2

SUMMARY:
Transcranial magnetic stimulation (TMS) is a noninvasive brain stimulation technique that is increasingly used for a growing number of research and clinical applications.Typically, this transient magnetic field is focally applied with a figure-of-eight coil that is carefully placed on the surface of the scalp over a targeted stimulation site. Patterned repetitive TMS (rTMS), such as theta burst stimulation (TBS) can produce long-lasting effects on neural activity and behavior beyond the stimulation period (Chou et al., 2015a; Fitzgerald et al., 2006). In general, high frequency (> 5 Hz) rTMS and its newer version, intermittent theta burst stimulation (iTBS), facilitate cortical excitability, whereas low frequency (about 1 Hz) rTMS and continuous theta burst stimulation contribute to opposite effects (Pascual-Leone et al., 2000; Huang et al., 2005; Wassermann and Zimmermann, 2012).Careful manipulation of the parameters comprising these patterned rTMS pulse trains can induce neuroplastic changes that resemble either long-term potentiation (LTP) or depression (Chen et al., 1997; Pascual-Leone et al., 1994). Early studies targeting the motor cortex helped elucidate which rTMS parameters promote particular responses and their neurophysiological underpinnings (Klomjai et al., 2015).

In recent years, rTMS has been closely investigated to evaluate its potential to modulate cognitive functions in Alzheimer'sdisease (AD) and mild cognitive impairment (MCI). As compared to conventional excitatory rTMS protocols, iTBS leads to comparable effects with similar number of pulses but considerable shorter duration and lower intensity of stimulation (Bakker et al., 2015; Rossi, Hallett, Rossini, Pascual-Leone, & Safety, 2009). Recent literature also suggest that TBS has lower rates of reported adverse event (AE) compared to rTMS (Najib & Horvath, 2014). Therefore, iTBS is assumed to modulate cognitive function in people with cognitive impairments.

DETAILED DESCRIPTION:
Visit 1: Informed Consent, Brain MRI/Neuropsychological Battery

Visit 2-11: (up to a week after visit 1) iTBS - or Sham-Treatment (10 sessions, 80% Resting Motor Threshold, 2s stimulation 8s inter-stimulus interval per train, 20 trains per block, 3 blocks per session with a 5-min break, 1 session per day)

Visit 12: (1 day or same day after visit 11) Functional Brain MRI/Neuropsychological Battery

Visit 13: (4 weeks after visit 11) Functional Brain MRI/Neuropsychological Battery

ELIGIBILITY:
Inclusion Criteria:

* normal visual acuity
* diagnosed with mild cognitive impairment or early dementia due to Alzheimer's disease (CDR = 0.5) by neurologists

Exclusion Criteria:

* (family) history of seizure attacks
* in intensive care
* history of drug/alcohol dependence
* assistants or students of the PI
* major systemic diseases concerning cognitive decline (e.g., cardiopulmonary failure, liver/renal failure, poor controlled DM, traumatic brain injury, stroke, or other neurodegenerative diseases)
* claustrophobia
* metal implants
* taking medication lowering the threshold of seizure attacks
* fear of using TMS
* with specific allergens
* pregnant or breastfeeding women

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in scores of any tests of the Neuropsychological Battery | Baseline, immediate post-iTBS, follow-up (4 weeks post-iTBS)
  WAIS-IV short-form, Word Sequence Learning Test, Benton Visual Retention Test, Color Trial Tests, 3-D Dimensional Constructional Test, Visual Confrontation Naming, Semantic Verbal Fluency Test, Stroop Color-Word Test

SECONDARY OUTCOMES:
Brain MRI | Baseline, immediate post-iTBS, follow-up (4 weeks post-iTBS)
  Change in white matter and brain activities at resting state at baseline compared to after iTBS stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Chun Kuan, MD, Principal Investigator — Taipei Medical University Shuang Ho Hospital
Locations (1):
- Shuang Ho Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang CC, Huang KY, Hsu JL, Hu CJ, Lu YH, Kuan YC. Effects of intermittent theta-burst stimulation on cognition and glymphatic system activity in mild cognitive impairment and very mild Alzheimer's disease: a randomized controlled trial. J Neuroeng Rehabil. 2025 Sep 26;22(1):195. doi: 10.1186/s12984-025-01738-1. PMID 41013466